CLINICAL TRIAL: NCT00179985
Title: The Impact of Implementing The Newborn Individualized Developmental Care & Assessment Program on the Developmental Sensitivity of Nurses Caring for Preterm Infants
Brief Title: The Impact of Implementing NIDCAP on the Developmental Sensitivity of Nurses Caring for Preterm Infants
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Susan M Horner, RNC, MS, Children's Memorial Hospital
Other Study IDs: IRB#2005-12423
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Infant, Premature Development
Keywords: Developmental Care; Neonatal Intensive Care Unit (NICU)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Training: Behavioral: Newborn Individualized Care and Assessment Program (NIDCAP)

SUMMARY:
The purpose of this study is to determine whether implementing the Newborn Individualized Developmental Care and Assessment Program increases NICU nurses' sensitivity in meeting the developmental care needs of preterm infants.

DETAILED DESCRIPTION:
Therapies that have brought about sharp decreases in neonatal mortality have not brought about similar decreases in neurodevelopmental morbidity for preterm infants. Developmentally supportive care is NICU (Neonatal Intensive Care Unit) care that seeks to optimize the developmental course and outcomes for preterm infants. In controlled trials, implementation of the Newborn Individualized Developmental Care and Assessment Program (NIDCAP) has been associated with with positive medical and neurobehavioral outcomes. The purpose of this study is to examine the impact of implementing the NIDCAP on the developmental sensitivity of nurses caring for preterm infants in a tertiary level NICU in a children's hospital in the midwest. The NIDCAP program consists of 1) structured behavioral observations which are conducted at regular intervals during the preterm infant's hospitalization, 2) written plans which outline specific, individualized interventions to address the infant's unique developmental needs which are updated following each observation, and 3) consultations with the infant's caregivers to articulate the infant's current needs and plan. A convenience sample of 32 NICU nurses will be observed during a routine caregiving episode with one preterm infant before and another preterm infant after the implementation of the NIDCAP program with preterm infants in the NICU. Following the observations, the nurse's developmental sensitivity will be scored using a standardized tool. The nurses' developmental sensitivity before the implementation of the NIDCAP program will be compared with their developmental sensitivity following NIDCAP implementation. Informed consent will be obtained from the nurses participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* be an RN,
* be an employee of the NICU at the study site,
* have completed the NICU nursing orientation at the study site,
* work at least 0.4 FTE in the NICU at the study site, and
* be observed while caring for a preterm infant born at less than or equal to 36 weeks gestation and at less than or equal to 1500 grams

Exclusion Criteria:

* Nurses will not be observed while caring for fullterm infants or preterm infants receiving heavy sedation or paralyzing medications.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: NICU Nurse
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2004-12; Primary Completion 2006-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pre-NIDCAP implementation and post-NIDCAP implementation, score on a tool designed to measure NICU nurses' developmental sensitivity. | Two years
  Measure NICU nurses' developmental sensitivity after training program

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Horner, RNC, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Neonatal Intensive Care Unit, Children's Memorial Hospital, Chicago, Illinois, United States